CLINICAL TRIAL: NCT03263325
Title: Evaluation of UDP-glucose as a Urinary Biomarker for Early Detection of Cardiac Surgery-associated Pediatric Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Douglas Atkinson, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00025852
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI Group: Patients developing AKI after surgery
  Interventions: Other: Discarded urine sample
- No AKI Group: Patients who do not develop AKI after surgery
  Interventions: Other: Discarded urine sample

INTERVENTIONS:
Other: Discarded urine sample — Collection of discarded urine during surgery and following surgery

SUMMARY:
Acute kidney injury (AKI) is common in children after cardiac surgery with a reported incidence of 20-40%. Pediatric AKI has been found to be associated with important short and long-term adverse outcomes.

A major challenge to management of AKI after cardiac surgery and cardiopulmonary bypass is the lack of early diagnostic markers. Current diagnostic criteria for AKI in children relies exclusively on elevation of serum creatinine concentration and oliguria. Both of these markers lack sensitivity and specificity, and result in delayed detection of kidney injury.

This study aims to determine if UDP-glucose can be used as a urinary biomarker to detect subclinical acute kidney injury following pediatric cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* less than or equal to 8 years of age
* scheduled for cardiac surgery

Exclusion Criteria:

* severe pre-existing renal insufficiency

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ≤ 8 years of age having cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
AKI | within 72 hours after surgery
  development of AKI

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Atkinson, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No